CLINICAL TRIAL: NCT05126498
Title: The Influence of the COVID-19 Pandemic on Surgical Patterns of Care in the Netherlands: a Prospective Nationwide Study
Brief Title: Influence of the COVID-19 Pandemic on Dutch Surgical Patterns of Care
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: COVIDsurgII01
Record Dates: First submitted 2021-11-16; First posted 2021-11-19 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: COVID-19
Keywords: surgery; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 2018: All surgically treated patients in the surgical audits for lung cancer surgery (DLCA-S), Upper gastrointestinal cancer surgery (DUCA), pancreatic cancer surgery (DPCA), hepatobiliary surgery (DHBA), colorectal cancer surgery (DCRA), hip fracture surgery (DHFA), aortic aneurysm surgery (DSAA), and bariatric surgery (DATO), from the participating hospitals in 2018
  Interventions: Other: no intervention
- Cohort 2019: All surgically treated patients in the surgical audits for lung cancer surgery (DLCA-S), Upper gastrointestinal cancer surgery (DUCA), pancreatic cancer surgery (DPCA), hepatobiliary surgery (DHBA), colorectal cancer surgery (DCRA), hip fracture surgery (DHFA), aortic aneurysm surgery (DSAA), and bariatric surgery (DATO), from the participating hospitals in 2019
  Interventions: Other: no intervention
- Cohort 2020: All surgically treated patients in the surgical audits for lung cancer surgery (DLCA-S), Upper gastrointestinal cancer surgery (DUCA), pancreatic cancer surgery (DPCA), hepatobiliary surgery (DHBA), colorectal cancer surgery (DCRA), hip fracture surgery (DHFA), aortic aneurysm surgery (DSAA), and bariatric surgery (DATO), from the participating hospitals in 2020
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention was applied

SUMMARY:
The aim of this study is to determine the impact of the COVID-19 pandemic on the Dutch surgical care, expressed as number of performed procedures, altered treatment plans, and surgical outcomes in the Netherlands during the year 2020.

DETAILED DESCRIPTION:
The aim of this study is to determine the impact of the COVID-19 pandemic on the Dutch surgical care, expressed as number of performed procedures, altered treatment plans, and surgical outcomes in the Netherlands during the year 2020. This was done by executing a nationwide prospective cohort study, under the name "Dutch COVIDsurg II Snapshot Study". This study was conducted in collaboration with the Dutch Institute of Clinical Auditing (DICA). For this study, the surgical audits for lung cancer surgery (DLCA-S), Upper gastrointestinal cancer surgery (DUCA), pancreatic cancer surgery (DPCA), hepatobiliary surgery (DHBA), colorectal cancer surgery (DCRA), hip fracture surgery (DHFA), aortic aneurysm surgery (DSAA), and bariatric surgery (DATO), were expanded with an additional COVID-19 survey, since August 2020. This survey focused on alterations in, or delay of treatment and diagnostics, perioperative outcomes, and specific COVID-19 related symptoms and complications during the COVID-19 pandemic. All academic-, general community-, teaching- and non-teaching hospitals in the Netherlands performing pulmonary, upper gastrointestinal, pancreatic, hepatobiliary, colorectal, hip fracture, aneurysmal or bariatric procedures were approached to participate in the Dutch COVIDSurg II Snapshot study. Patients who underwent surgery during the period January 1st 2018 until December 31st 2019, were included in the historical cohort. Patients who underwent a surgical procedure in the period January 1st 2020 until December 31st 2020 were included in the study group.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent pulmonary, upper gastrointestinal, pancreatic, hepatobiliary, colorectal, hip fracture, aneurysm or bariatric surgery
* Alle patients >18 years
* Patients undergoing surgery during the period January 1st 2018 until December 31st 2020
* Hospital that performs the surgery has to participate in the study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing pulmonary, upper gastrointestinal, pancreatic, hepatobiliary, colorectal, hip fracture, aneurysm or bariatric surgery in one of the participating hospitals during the period January 1st 2018 until December 31st 2020.
Sampling Method: Non-Probability Sample
Enrollment: 40296 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Number of performed surgical procedures | 2018-2020
  The data on surgical outcomes was collected through the database of the Dutch Institute for Clinical Auditing

SECONDARY OUTCOMES:
Length of hospital stay (days) | 2018-2020
  Data was collected through an additional COVID-19 survey and through the database of the Dutch Institute for Clinical Auditing
30-day hospital readmissions (percentage) | 2018-2020
  Data was collected through an additional COVID-19 survey and through the database of the Dutch Institute for Clinical Auditing
severe complications (Clavien-Dindo grade > 3A) | 2018-2020
  Severe complications are defined as Clavien-Dindo grading system
  Data was collected through an additional COVID-19 survey and through the database of the Dutch Institute for Clinical Auditing
ICU admission (percentage) | 2018-2020
  Data was collected through an additional COVID-19 survey and through the database of the Dutch Institute for Clinical Auditing
length of ICU stay (days) | 2018-2020
  Data was collected through an additional COVID-19 survey and through the database of the Dutch Institute for Clinical Auditing
mortality rate (percentage) | 2018-2020
  Data was collected through an additional COVID-19 survey and through the database of the Dutch Institute for Clinical Auditing
  Mortality is defined as mortality during hospital stay or within 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
no IPD will be shared